CLINICAL TRIAL: NCT00351520
Title: Phase 3, Clinical Trials of Drug Against Cutaneous Leishmaniasis
Brief Title: Efficacy Trial on Oral Miltefosine in Comparison With Glucantime in the Treatment of ACL Caused by L. Tropica
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: World Health Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGS05/97; WHO/EMRO
Record Dates: First submitted 2006-07-12; First posted 2006-07-13 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Cutaneous Leishmaniasis
Keywords: Anthoponotic Cutaneous leishmaniasis; Glucantime; Miltefosine
MeSH Terms: conditions — Leishmaniasis, Cutaneous

INTERVENTIONS:
Drug: Miltefose

SUMMARY:
Cutaneous leishmaniasis is a parasitic skin lesion caused by different species of Leishmania and transmitted by the bite of infected sand flies. Leishmaniasis is exist in 88 countries, pentavalent antimonials (sodium stibogluconate and meglumine antimoniate) have been used as a standard treatment for this disease for last 80 years. Pentavalent antimonials are only available as injectable, which is painful, toxic, not affordable and moreover is not always effective even sometimes with several courses of treatment. Many different modalities are used to treat the disease with little success. Miltefosine is drug and has recently been shown to be effective in the treatment cutaneous leishmaniasis in Colombia. The molecular mechanisms that contribute to this effectiveness are not clearly understood. Only a well designed, randomized clinical trial can precisely evaluate the efficacy of any therapeutic modalities in cutaneous leishmaniasis. In this study the efficacy of oral treatment of miltefosine 2.5 mg per Kg body weight for 4 weeks will be compared with standard treatment of intramuscular injections of 60 mg/kg/day glucantime for 2 weeks in ACL parasitologically proven patients. At 8 weeks after the initiation of the treatment any patient in the group who received miltefosine and has not responded to the treatment will be treated with the standard intramuscular injections of 60 mg/kg/day glucantime for 2 weeks. The clinical trial will be carried out according to the International approved GCP (Good Clinical Practice) guide lines.

DETAILED DESCRIPTION:
Leishmaniasis caused by at least 20 different species of Leishmania and transmitted by the bite of infected sand flies. Leishmaniasis is endemic in 88 countries, mostly developing ones. Leishmaniasis with an incidence rate of 1.5-2 million mostly cutaneous form, and 350 million population at risk is a major health problem in some endemic countries such as Iran which is endemic to cutaneous leishmaniasis (CL), both anthroponotic CL (ACL) caused by L. tropica and Zoonotic CL (ZCL) caused by L. major 1, 2. Pentavalent antimonials (sodium stibogluconate and meglumine antimoniate) have been used as standard treatment of leishmaniasis for about 80 years. Pentavalent antimonials are only parentrally available, which is painful, toxic, not affordable in most endemic areas and moreover is not always effective even sometimes with several courses of treatment, recently resistance of Leishmania to antimonials is reported. Other modalities such as physical, immunological, topical and systemic therapies are used with controversial results 3,4.

Miltefosine, is a phosphocholine analogue that affects cell-signaling pathways and membrane synthesis 5.

Almost all strains of mice are resistant to L. major and L. mexicana infection, in ressitant strain L. major infection induces a transient self healing lesion similar to human CL accompanies with a Th1 response but susceptible BALB/c mice infected with L. major induces a Th2 type immune response and the infection develop to a systemic form of disease similar to human Kala azar and eventually every mouse is succumed to the disease. Miltefosine has recently been shown to be effective in the treatment of visceral leishmaniasis (VL) caused by L. donovani and New World CL caused by L. vianna panamensis in Colombia 6-8. The results of an open-label, multicenteric, phase II trial of different doses of oral miltefosine (4 or 6 weeks) on patients with VL caused by L. donovani in India showed a cure rate of 95% (all 120 patients showed an initial parasitologic cure and relapsed was seen in only 6 patients) 6. In another randomized, open trial in India, VL patients received miltefosine orally (approximately 2.5 mg/kg daily for 28 days), or amphotericin B (1 mg/kg, every other day for 30 days) at the end of the treatment, parasitological cure rate was 100% and only 6% of the patients received miltefosien showed relapse by 6 months 7. Phase I-II of an open dose escalating trial of miltefosine against American CL in Colombia showed that oral miltefosine is safe and the cure rate was 66 and 94% for different doses 8. In a placebo-controlled trial of miltefosine in Colombia and Guatemala, American CL caused by L. v. panamensis was treated with miltfosine (2.5 mg/kg per day orally for 28 days), at the end of the teatment period, the per-protocol cure rates for miltefosine group was 91% and for placebo group was 38% 9.

The molecular mechanisms that contribute to the antileishmanial activity of miltefosine are not clearly understood but apparently the effect is not on immune response and macrophages since immunodefient mice such as SCID mice and other deficient mice are still susceptible to miltefosine action 10-12. It is shown that miltefosine induces nuclear DNA condensation and apoptosis-like death in L. donovani 12-14.

The controversy obsereved in the reports of the efficacy of different modalities for CL is mainly due to not considering the self healing nature of the disease in the design of the study. Factors such as variations in the susceptibility of different Leishmania species to the various drugs and differences in the criteria used to evaluate the efficacy of the drugs are important. Although no reliable report is available on the efficacy of glucantime in the treatment of ACL caused by L. tropica but surely the efficacy is very poor, and resistant of L. tropica to glucantime exist (manuscript submitted). Only with well designed, randomized clinical trial can precisely evaluate the efficacy of any therapeutic modalities in CL. In this study the efficacy of oral treatment of miltefosine 2.5 mg per Kg body weight for 4 weeks will be compared with standard treatment of intramuscular injections of 60 mg/kg/day glucantime for 2 weeks in ACL parasitologically proven patients. At 8 weeks after the initiation of the treatment any patient in the group who received miltefosine and has not responded to the treatment will be treated with the standard intramuscular injections of 60 mg/kg/day glucantime for 2 weeks. The clinical trial will be carried out according to GCP (Good Clinical Practice) guide lines.

Study area/setting: (Instructions: describe the area or setting where the study will be conducted. This description should cover the details relevant to the study topic) Study site: There are two sites of ACL with high incidence rate in Iran; one is Mashad, Khorasan and the second one is Bam, Kerman, the incidence rate of ACL in Bam is increasing after earthquake according to a recent survey which is currently underway. The trial will be carried out in either site with enough number of ACL patients, but also to complete the recruitment faster the trial could be carried out in both sites.

6.2 Study subjects: (Instructions: eligibility and exclusion criteria of the study subjects) I) Inclusion criteria:a) Parasitologically proven cases of CL based on positive smear and/or culture; b) Otherwise healthy subjects on the basis of medical history, physical examination and results of blood tests (complete blood count [CBC], liver function tests [LFT] and renal function tests [RFT]); c) Age 12-50 years; d) body weight more than 40 kilograms; e) willing to participate in the study and sign the informed consent (by the patient or his/her parent/guardian in case of younger than 18 years).

II) Exclusion criteria: a) Pregnant or lactating women; b) Duration of lesion more than 6 months; c) Number of lesions more than 5; d) Lesion(s) with bacterial supperinfection e) History of full course of standard treatment (antimonials); f) History of allergy to glucantime; g) Serious systemic illnesses (as judged by the physician); h) Participation in any drug trials in the last 60 days.

III) Withdrawal criteria:a) A serious adverse event occurs; b) Withdrawal of the consent.

Withdrawn cases will be treated according to the investigators opinion and beneficial of the patients at no cost. All withdrawn patients will be evaluated in final analysis (intent-to-treat analysis).

IV) Treatment: In this phase III, randomized open trial, subjects meeting inclusion criteria of the trial will be randomly allocated into two groups according to a randomization list. One group will be treated with 2.5 mg/kg body weight of oral miltefosine and the second group will be treated with intramuscular injections of 60 mg/kg/day glucantime for 2 weeks. The oral miltefosine tablets will be delivered to each patient on days 0, 7, 14 and 21. A written instruction sheet will be given to each included patient, and the patient will be instructed to contact the research team on appearance of symptoms suggesting severe side effects (intractable diarrhea and/or vomiting, symtoms of liver, kidney or hematopoietic system dysfunction. A copy of the randomization list with the codes will be kept at WR office. Eight weeks after the initiatin of the treatment, any patient who received oral miltefosine and has active lesion will be treated with intramuscular glucantime injections (60mg/kg/day for 14 days).

v) Follow-up: Every included patient will be visited at 1, 2, 3, 4, 8 and 24 weeks after the initiation of the treatment. The flow chart is attached.

6.3 Study design: (Instructions: mention the type of study design eg cross-sectional, case-control, intervention study, etc..) This trial is an open randomized clinical trial under GCP guide lines. The Center academic staffs are well qualified in training of GCP nationally and internationally, several clinical trials both in therapeutic and vaccine development have been completed by this group..

v) Follow-up: The patients will be visited at 1, 2, 3, 4, 8 and 24 weeks after the initiation of the treatment. The flow chart is attached.

6.3 Study design: (Instructions: mention the type of study design eg cross-sectional, case-control, intervention study, etc..) This study is a randomized, open clinical trial under GCP guide lines. The Center academic staff are well qualified in training of GCP nationally and internationally and have completed several clinical trials in both therapeutic and vaccine efficacy trials under GCP guide lines.

Cutaneous leishmaniasis: Skin lesions clinically suspicious and parasitologically proven by direct smear and/or culture. The study area is endemic for ACL but a portion of the Leishmania isolates will be used for charecterization and identification using monoclonal antibodies and PCR technique.

Clinical cure: The primary clinical efficacy parameter will be the complete re-epithelization of all lesions with disappearance of induration (with or without scar). No parasitological evaluation will be done on clinically cured lesions.

Clinical improvement: Reduction in the size of ulcer and induration. Treatment failure: No change or increase in the size of induration and ulcer. Relapse: Reappearance of the lesion at the site or periphery of the cured lesion will be considered as relapse.

Parasitological cure: Negative smear and culture at the end of the treatment and follow up period will be regarded as parasitological cure.

1. Leishmaniasis. Tropical Disease Research, Progress 1995-96. Thirteenth Programme Report, WHO, Geneva, 1997.
2. Dowlati Y. Cutaneous leishmaniasis: clinical aspect. Clin Dermatol 1996 ;14:425-31.
3. Dowlati Y. Treatment of cutaneous leishmaniasis (old world). Clin Dermatol 1996; 14:513-7.
4. Berman JD. Human leishmaniasis: clinical, diagnostic, and chemotherapeutic developments in.the last 10 years. Clin Inf Dis 1997; 24:684-703.
5. Schmidt-Ott R, Klenner T, Overath P, Aebischer T. Topical treatment with hexadecylphosphocholine (Miltex) efficiently reduces parasite burden in experimental cutaneous leishmaniasis. Trans R Soc Trop Med Hyg. 1999; 93(1):85-90
6. Jha TK., Sundras S, Thakur CP et al. Miltefosine, an oral agent, for the treatment of indian viceral leishmaniasis. N Engl J Med 1999; 341:1795-800.
7. Sundar S, Jha TK, Thakur CP, et al Oral miltefosine for Indian visceral leishmaniasis. N Engl J Med. 2002 ;347(22):1739-46.
8. Soto J, Toledo J, Gutierrez P, Nicholls RS, Padilla J, Engel J Fischer C, Voss A, Berman J, Treatment of American Cutaneous Leishmaniasis with Miltefosine, an Oral Agent. Clin. Infec. Dis. 2001;33:e57-e61
9. Soto J, Arana BA, Toledo J, et al. Miltefosine for new world cutaneous leishmaniasis Clin Infect Dis. 2004; 38(9):1266-72.
10. Leonard R, Hardy J, van Tienhoven G, et al. Randomized, double-blind, placebo-controlled, multicenter trial of 6% miltefosine solution, a topical chemotherapy in cutaneous metastases from breast cancer. J Clin Oncol. 2001; 19(21):4150-9.
11. Escobar P, Yardley V, Croft SL. Activities of Hexadecylphosphocholine (Miltefosine), AmBisome, and Sodium Stibogluconate (Pentostam) against Leishmania donovani in Immunodeficient scid Mice.Antimicrob.Agents and Chemotherapy, 2001;:, Vol. 45, No:61872-1875
12. Murray HW, Delph-Etienne S, Visceral Leishmanicidal Activity of Hexadecylphosphocholine (Miltefosine) in Mice Deficient in T Cells and Activated Macrophage Microbicidal Mechanisms. J. of Infec Dis. 2000;181:795-799
13. Paris C, Loiseau PM, Bories C, Breard J. Miltefosine induces apoptosis-like death in Leishmania donovani promastigotes. Antimicrob Agents Chemother. 2004; 48(3):852-9.
14. Verma NK, Dey CS. Possible mechanism of miltefosine-mediated death of Leishmania donovani. Antimicrob Agents Chemother. 2004; 48(8):3010-5.

ELIGIBILITY:
Inclusion Criteria:

* Parasitologically proven cases of CL based on positive smear and/or culture
* Otherwise healthy subjects on the basis of medical history, physical examination and results of blood test (if seemed necessary by the physician)
* Age 12-60 years
* Willing to participate in the study and sign the informed consent (by the patient or his/her parent/guardian in case of younger than 18 years).

Exclusion Criteria:

* Pregnant or lactating women
* Duration of lesion more than 6 months
* Number of lesions more than 4
* Ulcer size greater than 4 cm in their largest diameter
* History of full course of standard treatment (antimonials)
* History of allergy to Glucantime
* Serious systemic illnesses (as judged by the physician)
* Participation in any drug trials in the last 60 days

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 148 (Actual)
Dates: Start 2006-05; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Complete re-epithelization of the lesion(s)

SECONDARY OUTCOMES:
Improvement of the lesion(s)

CONTACTS AND LOCATIONS:
Overall Officials: Ali Khamesipour, Principal Investigator — Center for Research & Training in Skin Diseases & Leprosy, Tehran University of Medical Sciences
Locations (1):
- Ali Khamesipour, Bam, Kerman, Iran